CLINICAL TRIAL: NCT07164066
Title: A Comparative Analysis of Digital and Conventional Techniques for Prosthetic Rehabilitation of Edentulous Patients in Dubai.
Brief Title: Digital vs Conventional Prosthetic Rehab & Occlusal Analysis in Edentulous Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, May Al Janahi, Prosthodontist, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MBRU IRB-2024-374
Record Dates: First submitted 2025-07-28; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Edentulous Complete Denture Wearers; Dental Occlusion
Keywords: Edentulism; Digital Occlusal Analysis; Digital Dentures; Quality of life; Occlusion
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Dentures (Other): Participants will first receive conventionally fabricated dentures for both the upper and lower jaws. This set will be made using traditional techniques, including impressions, a custom tray, jaw relation recording, try-in, and final fitting. After the washout period, they will receive a second set created with the 3D-printed technique.
  Interventions: Device: Digital Occlusal Analysis Device
- Digital Dentures (Other): Complete dentures fabricated with digital workflow, including intraoral scanning, CAD/CAM design, and 3D printing, followed by clinical fitting.
  Interventions: Device: Digital Occlusal Analysis Device

INTERVENTIONS:
Device: Digital Occlusal Analysis Device — Computerized occlusal analysis performed using T-Scan and ModJaw devices to record occlusal contacts, timing, and force distribution during prosthesis fitting and function.

SUMMARY:
15 Patients requiring complete dentures will be recruited from Dubai Health. Each patient will receive two sets of dentures with a washout period between sets. Patients will remain blinded to the fabrication method used for each set.

* Group 1: Participants will first receive conventionally fabricated dentures for both the upper and lower jaws. This set will be made using traditional techniques, including impressions, a custom tray, jaw relation recording, try-in, and final fitting. After the washout period, they will receive a second set created with the 3D-printed technique.
* Group 2: Participants in this group will initially receive 3D-printed complete dentures through a digital workflow, which involves intraoral scanning, STL file export, digital design, design review with the patient, 3D printing, and final fitting. Following the washout period, they will then receive a conventionally fabricated set.

DETAILED DESCRIPTION:
To ensure randomization and reduce order effects, participants will be randomly assigned to Group 1 or Group 2 using a stratified randomization approach in Microsoft Excel. A computer-generated random number will determine group allocation, ensuring that both groups have a balanced distribution based on age, gender, and oral health status. The randomization process will assign participants to either receive conventional dentures first (Group 1) or digital dentures first (Group 2), with a washout period between treatments. By randomizing the sequence of denture delivery, this method will control for potential biases in patient-reported outcomes (OHIP-14, DSQ) and clinical assessments, ensuring that the order of treatment does not influence the study results.

The following outcomes will be analysed:

* Quality of life (Qol) through Oral Health Impact Profile (OHIP-14)
* Patient reported outcomes (PROMS)
* Occlusal analysis - through conventional and digital analysis devices
* Costs
* Number of appointments
* Time AccuracyOutcome Measures The primary outcome of this study is the assessment of occlusal analysis using conventional and digital techniques.

The secondary outcomes include:

* Oral health-related quality of life (OHRQoL), measured using the validated Oral Health Impact Profile (OHIP-14).
* Patient-reported outcomes (PROMs), assessed through the Denture Satisfaction Questionnaire (DSQ), evaluating comfort, aesthetics, speech, and functional satisfaction.
* Number of appointments, recorded as the total number of visits required for fabrication and delivery of both conventional and digital dentures.
* Time efficiency, measured by recording the clinical duration required for key stages such as impressions and final insertions.
* Denture accuracy, assessed through 3D scanning and superimposition analysis using Geomagic Control X software, quantifying deviations between the designed and fabricated dentures. Clinical evaluation of fit, retention, and stability will also be conducted using a standardized grading scale.
* Cost-effectiveness, evaluated using a model adapted from McKenna et al. (2014), where the total cost per patient is divided by the OHIP-14 improvement score to yield a cost per one-point improvement in quality of life. This is benchmarked against the minimally important difference (MID), defined as a 5-point improvement:

Cost-effectiveness ratio = Total cost per patient / OHIP-14 improvement score Benchmark = Cost per point × 5 This model provides a practical and meaningful way to interpret cost relative to patient-perceived improvement, supporting decisions on the integration of digital denture workflows.

The factors will be analyzed through a combination of validated patient-reported outcome measures, digital and conventional assessment techniques, and cost-effectiveness evaluations. Quality of life (QOL) will be assessed using the Oral Health Impact Profile (OHIP-14), a validated measure of oral health-related quality of life, while patient-reported outcomes (PROMS) will be evaluated using the Denture Satisfaction Questionnaire (DSQ) to assess patient satisfaction with comfort, aesthetics, speech, and function of conventional and digital dentures. Occlusal analysis will be conducted using both conventional and digital methods. Articulating paper will be used to assess occlusal contact number and occlusal contact area through visual inspection, while T-Scan and Modjaw will provide quantitative measurements of occlusal force distribution and balance between conventional and digitally fabricated dentures.

Cost, time efficiency, and accuracy will be compared between fabrication techniques. The total number of clinical visits and time spent on clinical and laboratory procedures will be recorded to determine workflow efficiency. A comparative cost analysis will evaluate direct expenses (materials, fabrication) and indirect costs (adjustments, remakes). Denture accuracy will be assessed through 3D scanning and superimposition analysis using Geomagic Control X software, quantifying deviations between the designed and fabricated dentures. Additionally, the fit, retention, and stability of the dentures will be evaluated using a standardized clinical grading scale. Additionally, Accuracy is defined as "the degree to which the result of a measurement, calculation, or specification conforms to the correct value or a standard" . In this study, accuracy pertains to how closely the fabricated complete dentures whether produced via digital or conventional methods match their intended designs and clinical specifications.

To evaluate this:

* Digital Dentures: The fabricated digital dentures will be scanned, and their STL files will be superimposed onto the original CAD designs using Geomagic Control X software. This process will generate a color-coded deviation map, quantifying discrepancies between the designed and fabricated dentures.
* Conventional Dentures: Similarly, conventional dentures will be digitized to obtain their STL files. These will be superimposed onto the corresponding digital designs using the same software and methodology. This allows for a direct, quantitative comparison of the accuracy between conventional and digital fabrication methods.
* Occlusal Accuracy: Occlusal accuracy will be assessed by evaluating the contact points and force distribution. For conventional dentures, articulating paper will be used to mark occlusal contacts, which will then be scanned to create digital models. These models will be superimposed onto the original designs using Geomagic Control X to analyze the location and distribution of occlusal contacts. For digital dentures, occlusal contacts will be assessed through the digital workflow, and similar superimposition techniques will be applied. This approach enables a comprehensive comparison of occlusal accuracy between the two fabrication methods.

By employing these standardized digital superimposition techniques, the study ensures a consistent and objective assessment of denture accuracy across both fabrication workflows, encompassing both the overall fit and occlusal parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adults above the age of eighteen years seeking replacement of missing teeth
* Edentulous patients 6 months after extraction of any teeth
* Males and Females

Exclusion Criteria:

* Temporomandibular Joint Disorders(TMD)
* Limited mouth opening
* History of Head and neck oncology
* Conditions- such as Psychiatric conditions and Neurological conditions-, such as Parkinson's disease and Alzheimer's

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Occlusal Force Distribution and Contact Accuracy | 12 months
  Quantitative assessment of occlusal contact number, area, timing, and force distribution in digital versus conventional complete dentures, measured using T-Scan and ModJaw systems, and validated against articulating paper marks.

SECONDARY OUTCOMES:
Oral Health-Related Quality of Life (OHRQoL) | 12 months
  Change in Oral Health Impact Profile (OHIP-14) total scores between digital and conventional dentures, reflecting impact on comfort, function, and psychosocial well-being.

OTHER OUTCOMES:
Clinical Time Efficiency | 12 months
  Mean chairside time (in minutes) required for each clinical step, including impressions, jaw relation recording, try-in, and final insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Elbishari, PhD, Principal Investigator — MBRU

IPD SHARING:
Plan to Share IPD: No
confidentiality

REFERENCES:
- [Background] McKenna G, Tsakos G, Burke F, Brocklehurst P. Managing an Ageing Population: Challenging Oral Epidemiology. Prim Dent J. 2020 Sep;9(3):14-17. doi: 10.1177/2050168420943063. PMID 32940594
- [Background] Muller F. Interventions for edentate elders--what is the evidence? Gerodontology. 2014 Feb;31 Suppl 1:44-51. doi: 10.1111/ger.12083. PMID 24446979
- [Background] Qadeer S, Kerstein R, Kim RJ, Huh JB, Shin SW. Relationship between articulation paper mark size and percentage of force measured with computerized occlusal analysis. J Adv Prosthodont. 2012 Feb;4(1):7-12. doi: 10.4047/jap.2012.4.1.7. Epub 2012 Feb 29. PMID 22439094
- [Background] Gerritsen AE, Allen PF, Witter DJ, Bronkhorst EM, Creugers NH. Tooth loss and oral health-related quality of life: a systematic review and meta-analysis. Health Qual Life Outcomes. 2010 Nov 5;8:126. doi: 10.1186/1477-7525-8-126. PMID 21050499